CLINICAL TRIAL: NCT00127647
Title: MK0476 Phase III Double-Blind Comparative Study - Allergic Rhinitis
Brief Title: An Approved Drug to Study a New Indication for Allergic Rhinitis (0476-327)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0476-327; MK0476-327; 2005_038
Record Dates: First submitted 2005-08-04; First posted 2005-08-08 (Estimated); Last update posted 2024-08-15 (Actual); Status verified 2022-01

CONDITIONS: Rhinitis, Allergic, Seasonal
MeSH Terms: conditions — Rhinitis, Allergic, Seasonal | interventions — montelukast

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (3):
- 1 (Experimental): montelukast sodium 5 mg, QD 2-weeks
  Interventions: Drug: montelukast sodium
- 2 (Experimental): montelukast sodium 10 mg QD 2-weeks
  Interventions: Drug: montelukast sodium
- 3 (Active Comparator): Pranlukast 225 mg BID 2-weeks
  Interventions: Drug: Comparator: pranlukast

INTERVENTIONS:
Drug: montelukast sodium — montelukast sodium; 5 mg, 10 mg QD 2-weeks.
  Other Names: MK0476; Singulair
  Arms: 1; 2
Drug: Comparator: pranlukast — Pranlukast 225 mg BID 2-weeks.
  Arms: 3

SUMMARY:
The purpose of this trial is to evaluate the efficacy and safety of an investigational drug in adult patients with allergic rhinitis.

ELIGIBILITY:
Inclusion Criteria:

* Japanese males and females with a 2-year documented history of seasonal allergic rhinitis symptoms and positive allergy testing (cedar, alder and/or cypress)

Exclusion Criteria:

* Patients with drug-induced rhinitis or non-allergic rhinitis, or patients who used anti-histamine drugs (within 2 weeks) before the start of the observation period

Ages: 15 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 1375 (Actual)
Dates: Start 2004-11; Primary Completion 2005-04 (Actual); Study Completion 2005-04 (Actual)

PRIMARY OUTCOMES:
Composite Nasal Symptom Score

SECONDARY OUTCOMES:
Daytime nasal symptom score, Nighttime nasal symptom score

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Result] Okubo K, Baba K. A double-blind non-inferiority clinical study of montelukast, a cysteinyl leukotriene receptor 1 antagonist, compared with pranlukast in patients with seasonal allergic rhinitis. Allergol Int. 2008 Dec;57(4):383-90. doi: 10.2332/allergolint.O-08-533. Epub 2008 Nov 1. PMID 18946234